CLINICAL TRIAL: NCT03032783
Title: A Two Step Approach to Allogeneic Hematopoietic Stem Cell Transplantation for Patients With Hematologic Malignancies-Increasing GVT Effects Without Increasing Toxicity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16D.606; JT 9551 (Other: JeffTrial Number)
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Whole-Body Irradiation; Cyclophosphamide; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (TBI, DLI, chemotherapy, HSCT) (Experimental): Patients undergo Total-Body Irradiation (TBI) twice daily on days -10 to -8 and and donor lymphocyte infusion (DLI) on day -6. Patients receive cyclophosphamide IV on days -3 and -2, tacrolimus IV beginning on day -1 and then orally at least 2 or 3 days prior to discharge with taper starting on day 42, and mycophenolate mofetil IV twice daily on days -1 to 28. Patients undergo Allogeneic Hematopoietic Stem Cell Transplantation on day 0.
  Interventions: Radiation: Total-Body Irradiation; Procedure: Donor Lymphocyte Infusion; Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Radiation: Total-Body Irradiation — Undergo Total Body Irradiation
  Other Names: Total Body Irradiation
Procedure: Donor Lymphocyte Infusion — Undergo Donor Lymphocyte Infusion
  Other Names: DLI; Donor Leukocyte Infusion
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 1-bis(2-chloroethyl)-amino-1-oxo-2-aza-5-oxaphosphoridin monohydrate; 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate; 6055-19-2; Carloxan; Ciclofosfamida; Ciclofosfamide; Clafen; CP monohydrate; CTX; Cycloblastin; Cyclophospham; Cyclophosphamid monohydrate; WR- 138719
Drug: Tacrolimus — Given IV
  Other Names: Fujimycin; 717865; 109581-93-3; Hecoria; Prograf; Protopic
Drug: Mycophenolate Mofetil — Given IV
  Other Names: 115007-34-6; 128794-94-5; 724229; Cellcept
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo Hematopoietic Stem Cell Transplantation
  Other Names: HSCT; HSC

SUMMARY:
This phase II trial studies the how well donor stem cell transplant works in treating patients with high risk hematologic malignancies. Giving total-body irradiation and chemotherapy before a donor stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. The donated stem cells may also replace the patient's immune cells and help destroy any remaining cancer cells.

DETAILED DESCRIPTION:
Primary Objective:

1. To assess 2 year probability of OS in high risk patients undergoing a myeloablative 2 step HSCT utilizing strategies to decrease relapse.

Secondary Objective:

1. To assess relapse incidence at 2 years post-HSCT of patients undergoing treatment on this protocol.
2. To assess regimen related toxicity and GVHD incidence at 2 years post-HSCT and severity in patients undergoing treatment on this protocol.
3. To assess the consistency and pace of engraftment.
4. To assess the pace of T cell and B cell immune recovery.

ELIGIBILITY:
Inclusion Criteria:

This treatment is for patients with high risk hematologic malignancies. High risk is defined as:

* Any patient with a hematologic malignancy in which allogeneic HSCT is pursued with the expectation of cure. Patients may have post-treatment residual disease, but the disease should be stable or minimally progressive and must be responsive to chemotherapy.
* Any patient with an untreated hematologic malignancy in which allogeneic HSCT is thought to be the sole or the best option for cure and in Patients without morphologic evidence of disease but with high risk features which would predict for relapsed despite remission at HSCT such as adverse cytogenetics, 3rd or greater CR, or failure to recover peripheral blood counts to normal ranges. While these patients do not have detectable disease by current methods, like all patients they have non-detectable disease which in their case is highly aggressive.
* Patients with uncommon diagnoses in which allogeneic HSCT is thought to be beneficial but are no comparable to the majority of patients on this protocol will not be counted in the statistical aims of the study and will be reported descriptively. The PI and at least one Co-I must document this exception in the study binder and the rationale for descriptive report. An example of a patient who may meet this criteria is someone with a malignancy that is an overlap of two different diagnoses or one whose malignancy is difficult to categorize. While this circumstance is expected to be rare, it will prevent patients with rare diagnoses to be treated off study and it will help maintain homogeneity of the study population.
* Patients must have one related donor who is HLA mismatched in the GVHD direction at two or more HLA loci (except as described below)
* Patients must have adequate organ function:
* Left Ventricular Ejection Fraction (LVEF) of ≥50%
* DLCO (adjusted for hemoglobin) ≥50% of predicted and FEV-1 ≥50%
* Adequate liver function as defined by a serum bilirubin ≤1.8, Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 x Upper Limit of Normal (ULN)
* Creatinine clearance of ≥ 60ml/min
* Karnofsky Performance Status (KPS) of ≥80% on the modified KPS tool (see Appendix)
* Patients must be willing to use contraception if they have childbearing potential
* Able to give informed consent
* Age ≥ 18 years of age

Exclusion Criteria:

* Modified KPS of <80%
* > 5 Comorbidity Points on the Hematopoietic Cell Transplant Co-Morbidity Index (HCT CI) (See Appendix) (Patients with greater than 5 points will be allowed for trial with approval of the PI and at least 1 Co-I not on the primary care team of the patient.) this is an adjustment to account for healthy patients who meet the spirit of this protocol but have histories that result in higher than HCT-CI 5 points. An example is a patient with a solid tumor malignancy in their remote history (adds 3 points to HCT-CI total) where the treatment for the malignancy occurred years to decades before and there has been complete recovery of toxicities.
* Human Immunodeficiency Virus (HIV) positive
* Active involvement of the central nervous system with malignancy
* Psychiatric disorder that would preclude patients from signing an informed consent
* Pregnancy, or unwillingness to use contraception if they have childbearing potential
* Patients with life expectancy of ≤ 6 months for reasons other than their underlying hematologic/oncologic disorder
* Alemtuzumab treatment within 8 weeks of HSCT admission
* ATG within 8 weeks of HSCT administration
* Inability to tolerate cyclophosphamide or undergo total body irradiation at the doses specified in the treatment plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | At two years
  Will be tested using an exact one-sided binomial test with alpha 0.05. The trial will be considered successful if the null hypothesis of 45% 2-year OS is rejected. In addition, the exact binomial 95% confidence interval for 2-year OS will be computed.

SECONDARY OUTCOMES:
Incidence of graft failure | Up to 2 years
  Should be less than 10%
Incidence of non-relapse mortality | Up to 2 years
  Should be less than 20% at 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Usama Gergis, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Thomas Jefferson University, Philadephia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/